CLINICAL TRIAL: NCT04942353
Title: Effects of Home-based Exercise Rehabilitation on Healthcare Utilization in HeartMate 3TM Patients: A Randomized Controlled Pilot Study (MOVE-LVAD)
Brief Title: Effects of Home-based Exercise Rehabilitation on Healthcare Utilization in HeartMate 3 Patients
Acronym: MOVE-LVAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Himabindu Vidula, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004656
Record Dates: First submitted 2021-06-17; First posted 2021-06-28 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure; Left Ventricular Dysfunction
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Exercise Rehabilitation (Experimental)
  Interventions: Behavioral: Home-based Exercise Rehabilitation.
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Home-based Exercise Rehabilitation. — Based on physical therapist or exercise physiologist assessment, subjects will receive an individualized exercise prescription for frequency, duration, and intensity of walking and strength training (including exercises using light-weight hand-weights and upper and lower body exercises using resistance bands). Research team will provide updated exercise prescription based on Garmin watch/Datos app activity data and Datos app data (including Borg scale).
  Arms: Home-based Exercise Rehabilitation
Behavioral: Usual Care — Patients receive a standardized recommendation to increase their walking activity to 30 minutes 5 days/week.
  Arms: Usual Care

SUMMARY:
To demonstrate that home-based exercise rehabilitation (HER) compared to usual care (UC) results in a significant reduction in healthcare utilization in HeartMate 3 (HM3) left ventricular assist device (LVAD) patients.(defined as rehospitalization, VAD Clinic visits, and ER visits during the 1st year after index discharge following LVAD implantation).

DETAILED DESCRIPTION:
HER Subjects:

Get Garmin activity watch (has its own smartphone app to be activated)*, Datos app Get resistance bands and light weights Exercise prescription: Initially by physical therapist prior to discharge home & updated every month.

UC Subjects:

Get Garmin activity watch (has its own smartphone app to be activated), Datos app Exercise prescription: Try to get to 30 min of exercise 5 days a week

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age on the date of randomization
* Patient implanted with a new HeartMate 3 LVAD at URMC
* Patients enrolling in the study at the time of index discharge home following new HM3 LVAD implantation will be evaluated by a HF cardiologist and physical therapist and will need to demonstrate ability to ambulate independently. Patients enrolling in the study after their index discharge home following HM3 LVAD implantation will be evaluated by a HF cardiologist or VAD Coordinator and will need to demonstrate ability to ambulate independently.
* Patient willing to participate in HER.
* Patient owns a smartphone with Internet connection.

Exclusion Criteria:

* Major comorbidities or limitations that may interfere with exercise training (including significant orthopedic/neurologic limitations, decompensated HF, uncontrolled arrhythmias, unstable angina).
* Patient with a life expectancy <12 months.
* Patient unwilling to sign the consent for participation.
* Patient unwilling or unable to cooperate with the study protocol
* Patient who does not anticipate being a resident of the area for the scheduled duration of the research study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Mean number of clinic visits | 1 year
  Healthcare utilization will be measured as the sum of all-cause rehospitalizations, outpatient VAD Clinic visits and emergency room visits room visits

SECONDARY OUTCOMES:
Mean number of days out of the hospital | 1 year
Mean change in the number of daily steps taken | 1 year
  Steps will be tracked using the Garmin watch. The Garmin watch uses Global Positioning System (GPS) tracking and an accelerometer to continuously monitor activity and provides data on average number of steps per day.
Mean change 6-minute walk distance | baseline to 1 year
Mean change in number of participants with improved quality of life | baseline to 1 year
  Quality of life will be measured using the Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12). The scale ranges from 12-70 with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No